CLINICAL TRIAL: NCT03553108
Title: A Phase 1, Randomised, Open-label, 4-Period Crossover Study to Develop an In Vitro-In Vivo Correlation for Olaparib Tablets in Subjects With Solid Tumors
Brief Title: A Study Using Olaparib Tablets for Subjects With Advanced Solid Tumours.
Acronym: IVIVC
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Collaborators: Iqvia Pty Ltd (Industry); Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: D0816C00024
Record Dates: First submitted 2018-05-14; First posted 2018-06-12 (Actual); Last update posted 2020-10-01 (Actual); Status verified 2020-09

CONDITIONS: Malignant Solid Tumor
Keywords: Solid Tumor

STUDY DESIGN:
Intervention Model Description: Protocol designed to evaluate one or more interventions for treating a disease, syndrome or condition
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Olaparib Treatment Sequence ABCD (Experimental): On Day 1 of each period, patients will receive a single dose of either Tablet A, B, C, or D, according to the randomization schedule. Serial blood samples for determination of olaparib in plasma will be collected for 72 hours.
  A - Olaparib Tablet 25 mg B - Olaparib Tablet 100 mg C - Olaparib Tablet 150 mg D - Olaparib Tablet 250 mg
  Interventions: Drug: Olaparib Treatment A; Drug: Olaparib Treatment B; Drug: Olaparib Treatment C; Drug: Olaparib Treatment D
- Olaparib Treatment Sequence BDAC (Experimental): On Day 1 of each period, patients will receive a single dose of either Tablet A, B, C, or D, according to the randomization schedule. Serial blood samples for determination of olaparib in plasma will be collected for 72 hours.
  B - Olaparib Tablet 100 mg D - Olaparib Tablet 250 mg A - Olaparib Tablet 25 mg C - Olaparib Tablet 150 mg
  Interventions: Drug: Olaparib Treatment A; Drug: Olaparib Treatment B; Drug: Olaparib Treatment C; Drug: Olaparib Treatment D
- Olaparib Treatment Sequence CADB (Experimental): On Day 1 of each period, patients will receive a single dose of either Tablet A, B, C, or D, according to the randomization schedule. Serial blood samples for determination of olaparib in plasma will be collected for 72 hours.
  C - Olaparib Tablet 150 mg A - Olaparib Tablet 25 mg D - Olaparib Tablet 250 mg B - Olaparib Tablet 100 mg
  Interventions: Drug: Olaparib Treatment A; Drug: Olaparib Treatment B; Drug: Olaparib Treatment C; Drug: Olaparib Treatment D
- Olaparib Treatment Sequence DCBA (Experimental): On Day 1 of each period, patients will receive a single dose of either Tablet A, B, C, or D, according to the randomization schedule. Serial blood samples for determination of olaparib in plasma will be collected for 72 hours.
  D - Olaparib Tablet 250 mg C - Olaparib Tablet 150 mg B - Olaparib Tablet 100 mg A - Olaparib Tablet 25 mg
  Interventions: Drug: Olaparib Treatment A; Drug: Olaparib Treatment B; Drug: Olaparib Treatment C; Drug: Olaparib Treatment D

INTERVENTIONS:
Drug: Olaparib Treatment A — Olaparib Tablet 25 mg
Drug: Olaparib Treatment B — Olaparib Tablet 100 mg
Drug: Olaparib Treatment C — Olaparib Tablet 150 mg
Drug: Olaparib Treatment D — Olaparib Tablet 250 mg

SUMMARY:
This is a phase 1 open label, 4 treatment, 4 sequence and 4 period crossover study in subjects with solid tumours no longer responding to, or eligible for standard therapies, and for whom there are no additional standard therapies likely to benefit the subject.

DETAILED DESCRIPTION:
The study is an open-label, randomised, 4-period, 4-sequence crossover pharmacokinetic study designed to generate in vivo PK data from tablet variants with different size/geometry and dose, to correlate with their corresponding in vitro dissolution profiles. The duration of each dosing period is 7 days including the washout period. Subjects will be randomised to a treatment sequence, following a balanced Latin Squares design. Twelve subjects who meet inclusion/exclusion criteria and have provided informed consent will be randomly assigned to the treatment sequences: ABCD, BDAC, CADB, or DCBA.

On Day 1 of each period, subjects will receive a single dose of either Treatment A, B, C, or D, according to the randomisation schedule. Serial blood samples for determination of olaparib in plasma will be collected for up to 72 hours.

Cancer subjects with advanced solid tumours are required for this study, as pre-clinical toxicology data preclude the use of olaparib in healthy volunteers. The olaparib doses chosen will deliver exposure at or below that which has been previously demonstrated to be acceptable and tolerated in cancer subjects.

ELIGIBILITY:
Inclusion Criteria:

1. Provision of informed consent prior to any study specific procedures.
2. Female or male subject, aged > 18 years.
3. Histologically or, where appropriate, cytologically confirmed malignant solid tumour refractory or resistant to standard therapy for which no suitable effective standard therapy is available and in the opinion of the investigator might benefit from olaparib therapy.
4. Subjects must have normal organ and bone marrow function measured within 28 days prior to administration of study treatment as defined below:

   * Haemoglobin ≥ 100 g/L with no blood transfusion in the past 28 days.
   * Absolute neutrophil count (ANC) ≥ 1.5 x 109/L.
   * Platelet count ≥ 100 x 109/L.
   * Total bilirubin ≤ 1.5 x institutional upper limit of normal (ULN).
   * Aspartate aminotransferase (AST) (Serum Glutamic Oxaloacetic Transaminase (SGOT)) / Alanine aminotransferase (ALT) (Serum Glutamic Pyruvate Transaminase (SGPT)) ≤ 2.5 x institutional upper limit of normal unless liver metastases are present in which case they must be ≤ 5x ULN.
   * Subjects must have creatinine clearance estimated of ≥51 mL/min using the Cockcroft-Gault equation or based on a 24 hour urine test:

   Estimated creatinine clearance =[(140-age [years]) x weight (kg) x 1.2] (x F)a serum creatinine (μmol/L) a where F=0.85 for females and F=1 for males
5. Eastern Cooperative Oncology Group (ECOG) performance status 0-1.
6. Subjects must have a life expectancy ≥ 16 weeks.
7. Postmenopausal or evidence of non-childbearing status for women of childbearing potential: negative urine or serum pregnancy test within 28 days of study treatment and confirmed prior to treatment on day 1.

8 Male subjects must use a condom during treatment and for 3 months after the last dose of olaparib when having sexual intercourse with a pregnant woman or with a woman of childbearing potential. Female partners of male subjects should also use a highly effective form of contraception if they are of childbearing potential.

9 Subjects must have normal GI tract anatomy and function (see exclusion criteria for specifics).

10 Subjects is willing and able to comply with the protocol for the duration of the study including undergoing treatment and scheduled visits and examinations.

Exclusion Criteria:

1. Involvement in the planning and/or conduct of the study (applies to both AstraZeneca staff and/or staff at the study site).
2. Previous randomisation in the present study.
3. Participation in another clinical study with an investigational product during the last 1 month.
4. Any previous treatment with a PARP inhibitor, including olaparib.
5. Resting ECG indicating uncontrolled, potentially reversible cardiac conditions, as judged by the investigator (e.g., unstable ischemia, uncontrolled symptomatic arrhythmia, congestive heart failure, QTcF prolongation > 500 ms, electrolyte disturbances, etc.) or subjects with congenital long QT syndrome.
6. Subjects receiving any systemic chemotherapy or radiotherapy (except for palliative reasons) within 3 weeks prior to study treatment.
7. Concomitant use of known strong CYP3A inhibitors (e.g. itraconazole, telithromycin, clarithromycin, protease inhibitors boosted with ritonavir or cobicistat, indinavir, saquinavir, nelfinavir, boceprevir, telaprevir) or moderate CYP3A inhibitors (e.g. ciprofloxacin, erythromycin, diltiazem, fluconazole, verapamil). The required washout period prior to starting olaparib is 2 weeks.
8. Concomitant use of known strong (e.g. phenobarbital, enzalutamide, phenytoin, rifampicin, rifabutin, rifapentine, carbamazepine, nevirapine and St John's Wort) or moderate CYP3A inducers (e.g. bosentan, efavirenz, modafinil). The required washout period prior to starting olaparib is 5 weeks for enzalutamide or phenobarbital and 3 weeks for other agents.
9. Persistent toxicities (Common Terminology Criteria for Adverse Event (CTCAE) > grade 2) caused by previous cancer therapy, excluding alopecia.
10. Subjects with myelodysplastic syndrome/acute myeloid leukaemia or with features suggestive of MDS/AML.
11. Subjects with symptomatic uncontrolled brain metastases. A scan to confirm the absence of brain metastases is not required. The subject can receive a stable dose of corticosteroids before and during the study as long as these were started at least 4 weeks prior to treatment. Subjects with spinal cord compression unless considered to have received definitive treatment for this and evidence of clinically stable disease for 28 days
12. Major surgery within 2 weeks of starting study treatment and subjects must have recovered from any effects of any major surgery.
13. Subjects considered a poor medical risk due to a serious, uncontrolled medical disorder, non-malignant systemic disease or active, uncontrolled infection. Examples include, but are not limited to, uncontrolled ventricular arrhythmia, recent (within 3 months) myocardial infarction, uncontrolled major seizure disorder, unstable spinal cord compression, superior vena cava syndrome, extensive interstitial bilateral lung disease on High Resolution Computed Tomography (HRCT) scan or any psychiatric disorder that prohibits obtaining informed consent.
14. Subjects unable to swallow orally administered medication and subjects with gastrointestinal disorders likely to interfere with absorption of the study medication including surgery on the upper GI tract and small bowel, malabsorptive disorders, inflammatory bowel disease, GI motility disorders, chronic diarrhea (more than 3 loose bowel movements per day) chronic constipation (no bowel movement for more than two days), recent (in last week) vomiting.
15. Pregnant or breastfeeding women.
16. Immunocompromised subjects, e.g., subjects who are known to be serologically positive for human immunodeficiency virus (HIV).
17. Subjects with a known hypersensitivity to olaparib or any of the excipients of the product.
18. Subjects with known active hepatitis (i.e. Hepatitis B or C) due to risk of transmitting the infection through blood or other body fluids.
19. Previous allogenic bone marrow transplant or double umbilical cord blood transplantation (dUCBT).

Ages: 18 Years to 130 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2018-05-16 (Actual); Primary Completion 2019-03-12 (Actual); Study Completion 2020-07-01 (Actual)

PRIMARY OUTCOMES:
%PECmax | 0 to 72 hours
  Percent prediction error for Cmax
%PEAUC | 0 to 72 hours
  Percent prediction error for AUC

SECONDARY OUTCOMES:
Maximum plasma concentration (Cmax) obtained directly from the observed concentration versus time data. | Blood samples will be taken at the following sampling times: Pre-dose, 30 min, 1 hr, 1.5 hr, 2 hr, 2.5 hr, 3 hr, 4 hr, 6 hr, 8 hr, 12 hr (Day 1), 24 hr (Day2), 48 hr (Day 3), and 72 hr (Day 4). After each dosing at each of the 4 treatment cycles.
  Evaluation of the PK parameters for the different Olaparib tablet variants.
Time to maximum plasma concentration (tmax) obtained directly from the observed concentration versus time data. | Blood samples will be taken at the following sampling times: Pre-dose, 30 min, 1 hr, 1.5 hr, 2 hr, 2.5 hr, 3 hr, 4 hr, 6 hr, 8 hr, 12 hr (Day 1), 24 hr (Day2), 48 hr (Day 3), and 72 hr (Day 4). After each dosing at each of the 4 treatment cycles.
  Evaluation of the PK parameters for the different Olaparib tablet variants.
Area under the plasma concentration-time curve from zero to the time of the last measurable concentration (AUC(0-t)) calculated by linear up/log down trapezoidal summation. | Blood samples will be taken at the following sampling times: Pre-dose, 30 min, 1 hr, 1.5 hr, 2 hr, 2.5 hr, 3 hr, 4 hr, 6 hr, 8 hr, 12 hr (Day 1), 24 hr (Day2), 48 hr (Day 3), and 72 hr (Day 4). After each dosing at each of the 4 treatment cycles.
  Evaluation of the PK parameters for the different Olaparib tablet variants.
Area under the plasma concentration time curve from zero (pre-dose) extrapolated to infinity (AUC) | Blood samples will be taken at the following sampling times: Pre-dose, 30 min, 1 hr, 1.5 hr, 2 hr, 2.5 hr, 3 hr, 4 hr, 6 hr, 8 hr, 12 hr (Day 1), 24 hr (Day2), 48 hr (Day 3), and 72 hr (Day 4). After each dosing at each of the 4 treatment cycles.
  Evaluation of the PK parameters for the different Olaparib tablet variants. calculated by linear up/log down trapezoidal summation and extrapolated to infinity by addition of the last quantifiable concentration divided by the terminal rate constant: AUC(0-t) + Clast/λz.
Apparent plasma clearance (CL/F). | Blood samples will be taken at the following sampling times: Pre-dose, 30 min, 1 hr, 1.5 hr, 2 hr, 2.5 hr, 3 hr, 4 hr, 6 hr, 8 hr, 12 hr (Day 1), 24 hr (Day2), 48 hr (Day 3), and 72 hr (Day 4). After each dosing at each of the 4 treatment cycles.
  Evaluation of the PK parameters for the different Olaparib tablet variants.
Terminal half-life (t½). Visual assessment will be used to identify the terminal linear phase of the concentration-time profile. | Blood samples will be taken at the following sampling times: Pre-dose, 30 min, 1 hr, 1.5 hr, 2 hr, 2.5 hr, 3 hr, 4 hr, 6 hr, 8 hr, 12 hr (Day 1), 24 hr (Day2), 48 hr (Day 3), and 72 hr (Day 4). After each dosing at each of the 4 treatment cycles.
  Evaluation of the PK parameters for the different Olaparib tablet variants.
Apparent volume of distribution (Vz/F). | Blood samples will be taken at the following sampling times: Pre-dose, 30 min, 1 hr, 1.5 hr, 2 hr, 2.5 hr, 3 hr, 4 hr, 6 hr, 8 hr, 12 hr (Day 1), 24 hr (Day2), 48 hr (Day 3), and 72 hr (Day 4). After each dosing at each of the 4 treatment cycles.
  Evaluation of the PK parameters for the different Olaparib tablet variants.
Terminal rate constant (λz) estimated by log-linear least squares regression of the terminal part of the concentration-time curve. | Blood samples will be taken at the following sampling times: Pre-dose, 30 min, 1 hr, 1.5 hr, 2 hr, 2.5 hr, 3 hr, 4 hr, 6 hr, 8 hr, 12 hr (Day 1), 24 hr (Day2), 48 hr (Day 3), and 72 hr (Day 4). After each dosing at each of the 4 treatment cycles.
  Evaluation of the PK parameters for the different Olaparib tablet variants.

CONTACTS AND LOCATIONS:
Overall Officials: Kevin Punie, Principal Investigator — Universitaire Aiekenhuizen Leuven; Luc Dirix, Principal Investigator — GZA Ziekenhuizen; Guy Jerusalem, Principal Investigator — Centre Hospitalier Universitaire de Liege
Locations (3):
- Belgium (3):
  - Research Site, Leuven
  - Research Site, Liège
  - Research Site, Wilrijk

IPD SHARING:
Plan to Share IPD: No
Study team has decided that IPD would not be shared at this moment.